CLINICAL TRIAL: NCT03874650
Title: Mood, Activity Participation, and Leisure Engagement Satisfaction (MAPLES): A Pilot Feasibility Study for Low Mood in Acquired Brain Injury
Brief Title: MAPLES Pilot Study for Low Mood in ABI
Acronym: MAPLES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Tom Manly, Programme Leader, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2026112018
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Acquired Brain Injury; Depression
Keywords: acquired brain injury; traumatic brain injury; depression; rehabilitation; executive function
MeSH Terms: conditions — Brain Injuries; Depression; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Given that this is a psychological assessment, it is not possible to mask the participant, care provider, or investigator. Hence, only the outcomes assessor will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Activity Planning Group (Experimental): Those in the Activity Planning group receive training and practice in identifying realistic and safe activities in everyday life that may be enjoyable or rewarding to complete. They gain practice in scheduling activities and identifying and overcoming barriers to completion, such as memory problems, avoidance, sticking to habitual patterns and physical and transport issues.
  The intervention will consist of weekly 1 hour group sessions over 8 weeks, as below:
  Introduction to Group Therapy Identifying Enjoyable Activities The Automatic Pilot and Planning Pleasurable Activities Goal Review and Balancing Enjoyable and Routine Activities Identifying Solutions to Goal Attainment Increasing Mastery and Managing Fatigue Active Approaches to Engagement Relapse Prevention
  Interventions: Behavioral: Activity Planning Group
- Activity Engagement Group (Experimental): Individuals randomised to this arm will meet weekly for 8 weeks for 1 hour and engage in various potentially rewarding and meaningful social activities such as board games, crafting, and puzzles. Participants in this group will not receive specific training on activity scheduling or overcoming barriers to activity participation. Rather the aim is that participants gain experience of positive reinforcement from the activities and that this explicitly or implicitly challenges potentially negative predictions about such situations and encourages generalised increases in positive activity beyond the group setting. The group will cover activities such as board games, t-shirt making, puzzles, painting, "pub quizzes", figurine painting, origami/paper-craft, and clay sculptures.
  Interventions: Behavioral: Activity Engagement Group
- Waitlist Group (Placebo Comparator): In consenting to the study, individuals understand that access to groups cannot always be immediate. In the design we take advantage of this by completing the outcome measures before and after an 8-week period in participants randomized to this condition. We do not ask participants in any condition to discontinue any clinical services that they currently receive, hence the waitlist forms a treatment as usual control arm against which to judge and effects of the two groups. At the end of the waitlist the participants will be invited to take part in the Activity Planning or Activity Engagement Group depending upon their initial randomisation..
  Interventions: Behavioral: Waitlist Group

INTERVENTIONS:
Behavioral: Activity Planning Group — Participants in this group will receive 8 1-hour sessions of Behavioural Activation combined with select Goal Management Training strategies over the course of 8 weeks.
  Arms: Activity Planning Group
Behavioral: Activity Engagement Group — Participants in this group will attend 8 1-hour sessions of various social activities such as board games and puzzles.
  Arms: Activity Engagement Group
Behavioral: Waitlist Group — Participants in this group will continue on their care as usual before being re-randomised into either the Activity Planning Group or Activity Engagement Group after 8 weeks.
  Arms: Waitlist Group

SUMMARY:
Low mood and depression are common following acquired brain injury (ABI). There is a lack evidence on effective treatments in ABI. Behavioural Activation (BA) is a potentially valuable option. People with low mood can have problems imagining, planning and engaging in positive activities, or avoid activities due to fear of negative consequences. This can reduce positive reinforcement, further lowering mood. BA aims to reverse this cycle by encouraging individuals to engage in enjoyable activities. Despite its simplicity, it has been as effective as "talking therapies" and mood medication in non-ABI populations. Its simplicity may be particularly helpful in ABI where cognitive problems can form additional barriers to activity engagement.

This study will examine two ways to increase activity levels and improve mood. The first (Activity Engagement Group) is a social group run once a week for 8 weeks in which ABI participants will be encouraged to engage in games, crafts and discussion. The aim is that members gain direct positive reinforcement and may challenge fears such that activity levels could be maintained and mood enhanced after the group ends.

The second approach (Activity Planning Group), again an 8-week group, is to help participants identify, plan and schedule positive activities. The group will include discussion on identifying and overcoming problems in planning activities. Again, the hope is that training skills in planning and scheduling will generalise beyond the group.

The primary purpose is to examine the practicality, feasibility, and acceptability of the two approaches in ABI. A secondary purpose is to evaluate whether either group leads to improvements in activity levels and mood compared to a waitlist group. Individuals will be randomised to the Activity Engagement, Activity Planning Group or the 8-week Waitlist group. All will complete measures of activity levels and mood. At the end of the groups, these measures will be repeated. Waitlist participants will then be re-randomised to either the Activity Engagement Group or the Activity Planning Group.

Recruitment rates, drop out rates, and exit interviews will be used to assess feasibility and how meaningful or valuable participants found the groups. Comparison of measures will provide some indication of whether the groups are associated with improvements compared to those waitlisted. To establish whether any benefits last, all participants will repeat the measures 1 month after the groups end.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of an acquired brain injury (e.g., traumatic brain injury, stroke)
2. Speak and comprehend English
3. Are a minimum of 3 months post-acquired brain injury
4. Are identified as having low mood. Low mood will be identified by either:

   1. A score of at least 7 on the depression subscale of the Hospital Anxiety and Depression Scale, indicating clinically significant levels of depression, or
   2. Clinicians have identified that a client has low mood (i.e., through their own administration of the HADS within the past 3 months, through clinical interview determining that the client has low mood or would benefit emotionally from increased activity level)

Exclusion Criteria:

1. Are incapable of attending to and/or understanding the intervention materials (i.e., severe cognitive disability)
2. Have a diagnosis of dementia or other neurodegenerative disorder
3. Unstable psychotropic medication (i.e., have recently started/recently changed medications)
4. Are actively suicidal (i.e., have attempted suicide in the past 3 months, currently self-harm, and/or have a concrete plan to attempt suicide in the future, as identified by recurring clinician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Behavioural Activation for Depression Scale (BADS; Kanter et al., 2007) | Baseline, 1 week post-intervention, 1 month post-intervention
  This measure assesses changes in activity level related to depression. It consists of four subscales, Activation (engaging in meaningful activities) and Avoidance/Rumination (avoiding meaningful activities), Work/School impairment, and Social Impairment. To score the BADS, items from all scales other than the Activation scale are reverse-coded and then all items are summed. To score the subscales, no items are reverse-coded. For the total scale, higher scores represent increased activation, while for the Social Impairment subscale, higher scores represent increased social impairment. The minimum possible score on the BADS is 0, while the maximum possible is 150.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983) | Baseline, 1 week post-intervention, 1 month post-intervention
  This measure assesses levels of depression (subscale 1) and anxiety (subscale 2) in clinical settings. Each subscale is scored independently. On each subscale, each item is summed with no reverse-coded items. Greater scores on either subscale represent greater depression or anxiety. The minimum possible score on each subscale is 0, while the maximum possible score on each subscale is 21. Higher scores indicate greater depression and anxiety.
Behavioural Inhibition/Behavioural Activation Scales (BIS/BAS; Carver & White 1994) | Baseline, 1 week post-intervention, 1 month post-intervention
  This measures assesses individual disposition toward avoiding and engaging in activities. The BIS/BAS has three behavioural activation (BA) subscales, and only one subscale assesses behavioural inhibition (BI). The BA subscales are Drive, Fun Seeking, and Reward Responsiveness. All items except for two are reverse coded. Four items are filler questions and are not used for the subscale scores. Once the appropriate questions are reverse coded, each subscale is summed to get the respective subscale scores. The minimum score on BA Drive is 4, maximum 16. Higher scores indicate greater drive to engage. The minimum score on the BA Fun Seeking subscale is 4, maximum 16. Higher scores indicate greater fun seeking. The minimum score on the BA Reward Responsiveness subscale is 5, maximum 20. Higher scores indicate greater reward responsiveness.The minimum score on the BI subscale is 7, maximum 28. Greater scores indicate greater behavioural inhibition.
Intolerance of Uncertainty Scale-Short Form (IUS-SF; Carleton, Norton, & Asmundson) | Baseline, 1 week post-intervention, 1 month post-intervention
  This measure assesses the degree to which an individual is bothered by uncertainty. The IUS-SF has two subscales, Prospective Anxiety (concerns about the future), and Inhibitory (concerns prevent one from doing things). The items on the subscale are summed. No items are reverse-coded. A total score can be produced from combining two subscales. The minimum score on the Prospective Anxiety subscale is 5, maximum 25. Greater scores indicate greater prospective anxiety. The minimum score on the Inhibitory Anxiety subscale is 7, maximum 35. Greater scores indicate greater inhibitory anxiety.
Impact of Events Scale-Revised (IES-R, Weiss, 2007) | Baseline, 1 week post-intervention, 1 month post-intervention
  This measure assesses acute and routine life stress. The IES-R has three subscales, Avoidance (not thinking of stressful events), Intrusion (whether memories of stressful events occur) and Hyperarousal (The degree to which stressful events cause somatic symptoms). No items are reverse-coded. Although each subscale can produce a score, typically the total score is summed to determine the level of impact a stressful event has had on an individual. The items on the subscale are summed, ranging from 0 to 88. Scores 24 or higher indicate cause for clinical concern, 33 represents a probably diagnosis of post-traumatic stress disorder, and 37 is high enough to suppress immune function (i.e., severe clinical concern).
Brain Injury Rehabilitation Trust Motivation Questionnaire-Self (BMQ-S) | Baseline, 1 week post-intervention, 1 month post-intervention
  This measure assesses difficulties with overall motivation after brain injury. The scale has no subscales, and has 15 reverse-scored items. Once the appropriate questions are reverse scored, all items are summed to generate a total score. The minimum possible score is 34, maximum 136. Greater scores indicate greater difficulties with motivation.
Modified Outcome Measure - Participation Objective, Participation Subjective (MOM-POPS, Brown et al., 2004) | Baseline, 1 week post-intervention, 1 month post-intervention
  This is a modified measure of desired and actual participation in home and community activities. The scale contains 3 items, asking participants to rate their involvement in, frequency of, and importance of household, occupational, and social activities. Participants are then asked to check off which activities they have engaged in the past week, such as cleaning the house, made social arrangements, attended religious services, etc. Each item is scored individually, hence there is no score total. The first 3 items represent desired participation in daily activities, and the final item represents actual participation.
Sense of Control Scale (SCS; Lachman & Weaver, 1998a, 1998b) | Baseline, 1 week post-intervention, 1 month post-intervention
  This measure assesses perceived ability to exert control over one's life. It consists of two subscales, Perceived Constraints (i.e., whether there are barriers to control) and Perceived Mastery (one's subjective belief about their competency in one's life). All items on the perceived constraints scale are reverse coded. Each subscale is summed and interpreted independently. The minimum possible score on the Perceived Constraints scale is 8, maximum 56. Greater scores indicate more constraints.The minimum possible score on the Perceived Mastery subscale is 4, maximum 28. Greater scores indicate greater mastery.
Motivation for Traumatic Brain Injury Rehabilitation Questionnaire (MOT-Q; Chervinsky et al., 1998) | Baseline, 1 week post-intervention, 1 month post-intervention
  This scale assesses level of motivation toward rehabilitation-related activities in traumatic brain injury. It consists of 4 subscales, Lack of Denial (good insight), Interest in Rehabilitation, Lack of Anger, and Reliance on Professional Help. The MOT-Q uses a 5-point Likert scale from -2 to +2. The scale contains 19 reverse coded items. Each subscale is totaled separately, and can be added together to produce a total score. Higher scores indicate greater motivation for rehabilitation. Total scores can range from -62 to +62. The Lack of Denial subscale ranges from -16 to +16, with higher scores indicating better insight. The Interest in Rehabilitation subscale ranges from -14 to +14, with greater scores indicating greater interest. The Lack of Anger scubscale ranges from -20 to +20, with higher scores indicating lower anger. The Reliance on Professional Help subscale ranges from -12 to +12, with higher scores indicating greater reliance.
Credibility/Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000) | Baseline only
  This scale assesses participant expectations of treatment outcome and perceived credibility of treatment. It consists of 6 items. The first 4 items reflect what one think about the intervention, and the last 2 items evaluate how one feels about the intervention. This measure has two factors, Credibility and Expectancy. The Credibility subscale ranges from 3 to 27. Two items on the Expectancy subscale are perecentage based (0 to 100%) and the third item is Likert based from 1 to 9. Typically, items are evaluated individually rather than produce a scale total
Snaith Hamilton Pleasure Scale (SHAPS; Snaith et al., 1995) | Baseline, 1 week post-intervention, 1 month post-intervention
  This scale assesses level of ability to experience pleasure in day-to-day activities. It consists on 14 items, with 7 items reverse coded. Greater scores indicate greater ability to experience pleasure in daily activities. Once the appropriate items are reverse-coded, all items are summed. The minimum possible score is 14, maximum 56.
Fatigue Severity Scale (FSS; Krupp et al., 1989) | Baseline, 1 week post-intervention, 1 month post-intervention
  This scale assess overall levels of fatigues in patient populations within the past week. It consists of 7 Likert-rated items and one visual analogue scale for participants to rate overall fatigue. Greater scores indicate higher levels of fatigue. The minimum possible score is 7, maximum 49.
Generalized Anxiety Disorder-7 (GAD-7; Spitzer et al., 2006) | Baseline, 1 week post-intervention, 1 month post-intervention
  This scale measures symptoms of generalized anxiety disorder such as excessive worry and irritability, over the past two weeks. It consists of 8 items, with greater scores indicating greater anxiety. The minimum possible score is 0, and the highest possible score is 24.
Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001) | Baseline, 1 week post-intervention, 1 month post-intervention
  This scale measures symptoms of depression such as poor appetite or difficulties concentrating, over the past two weeks. It consists of 8 items, with greater scores indicating greater anxiety. The minimum possible score is 0, and the highest possible score is 24.
Verbal and Spatial Reasoning Test (VESPAR; Langdon & Warrington, 1995) | Baseline only
  This neuropsychological assessment measures fluid intelligence in neurological patients. It consists of 3 verbal and 3 spatial reasoning tasks, designed to calculate an individual's IQ.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Manly, PhD, Principal Investigator — University of Cambridge
Locations (2):
- United Kingdom (2):
  - Cambridgeshire Community Services, Cambridge, Cambs
  - Cambridge University Hospitals NHS Trust, Cambridge

IPD SHARING:
Plan to Share IPD: Yes
Only anonymised participant data from the study will be made accessible to other researchers upon publication of the study results. All data from all measures, including the questionnaires and qualitative interviews, will be made available once the study is completed. As we intend to publish the study as an open access article, all anonymised data will be available potentially indefinitely.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The study protocol and statistical analysis plan will be made available upon registration of the trial, along with publication of the trial protocol. This is expected to occur before May 2019. Analytic code will be made available upon publication of the study results, approximately 1 year following the completion of the trial (February 2022).
Access Criteria: The study protocol, statistical analysis plan, and analytic code will be available to any interested party.

REFERENCES:
- [Background] Brown M, Dijkers MP, Gordon WA, Ashman T, Charatz H, Cheng Z. Participation objective, participation subjective: a measure of participation combining outsider and insider perspectives. J Head Trauma Rehabil. 2004 Nov-Dec;19(6):459-81. doi: 10.1097/00001199-200411000-00004. PMID 15602309
- [Background] Carleton RN, Norton MA, Asmundson GJ. Fearing the unknown: a short version of the Intolerance of Uncertainty Scale. J Anxiety Disord. 2007;21(1):105-17. doi: 10.1016/j.janxdis.2006.03.014. Epub 2006 May 2. PMID 16647833
- [Background] Carver CS, White TL. Behavioural inhibition, behavioural activation, and affective responses to impending reward and punishment: The BIS/BAS scales. J Pers Soc Psychol, 67, 319-333, 1994.
- [Background] Cattelani R, Zettin M, Zoccolotti P. Rehabilitation treatments for adults with behavioral and psychosocial disorders following acquired brain injury: a systematic review. Neuropsychol Rev. 2010 Mar;20(1):52-85. doi: 10.1007/s11065-009-9125-y. Epub 2010 Feb 9. PMID 20143264
- [Background] Dimidjian S, Hollon SD, Dobson KS, Schmaling KB, Kohlenberg RJ, Addis ME, Gallop R, McGlinchey JB, Markley DK, Gollan JK, Atkins DC, Dunner DL, Jacobson NS. Randomized trial of behavioral activation, cognitive therapy, and antidepressant medication in the acute treatment of adults with major depression. J Consult Clin Psychol. 2006 Aug;74(4):658-70. doi: 10.1037/0022-006X.74.4.658. PMID 16881773
- [Background] Fazel S, Wolf A, Pillas D, Lichtenstein P, Langstrom N. Suicide, fatal injuries, and other causes of premature mortality in patients with traumatic brain injury: a 41-year Swedish population study. JAMA Psychiatry. 2014 Mar;71(3):326-33. doi: 10.1001/jamapsychiatry.2013.3935. PMID 24430827
- [Background] Hyder AA, Wunderlich CA, Puvanachandra P, Gururaj G, Kobusingye OC. The impact of traumatic brain injuries: a global perspective. NeuroRehabilitation. 2007;22(5):341-53. PMID 18162698
- [Background] Jorge RE, Robinson RG, Moser D, Tateno A, Crespo-Facorro B, Arndt S. Major depression following traumatic brain injury. Arch Gen Psychiatry. 2004 Jan;61(1):42-50. doi: 10.1001/archpsyc.61.1.42. PMID 14706943
- [Background] Kanter JW, Manos RC, Bowe WM, Baruch DE, Busch AM, Rusch LC. What is behavioral activation? A review of the empirical literature. Clin Psychol Rev. 2010 Aug;30(6):608-20. doi: 10.1016/j.cpr.2010.04.001. PMID 20677369
- [Background] Raes F, Hoes D, Van Gucht D, Kanter JW, Hermans D. The Dutch version of the Behavioral Activation for Depression Scale (BADS): psychometric properties and factor structure. J Behav Ther Exp Psychiatry. 2010 Sep;41(3):246-50. doi: 10.1016/j.jbtep.2010.02.001. Epub 2010 Feb 10. PMID 20167307
- [Background] Lachman ME, Weaver SL. Sociodemographic variations in the sense of control by domain: findings from the MacArthur studies of midlife. Psychol Aging. 1998 Dec;13(4):553-62. doi: 10.1037//0882-7974.13.4.553. PMID 9883456
- [Background] Lachman ME, Weaver SL. The sense of control as a moderator of social class differences in health and well-being. J Pers Soc Psychol. 1998 Mar;74(3):763-73. doi: 10.1037//0022-3514.74.3.763. PMID 9523418
- [Background] Levine B, Robertson IH, Clare L, Carter G, Hong J, Wilson BA, Duncan J, Stuss DT. Rehabilitation of executive functioning: an experimental-clinical validation of goal management training. J Int Neuropsychol Soc. 2000 Mar;6(3):299-312. doi: 10.1017/s1355617700633052. PMID 10824502
- [Background] Levine B, Schweizer TA, O'Connor C, Turner G, Gillingham S, Stuss DT, Manly T, Robertson IH. Rehabilitation of executive functioning in patients with frontal lobe brain damage with goal management training. Front Hum Neurosci. 2011 Feb 17;5:9. doi: 10.3389/fnhum.2011.00009. eCollection 2011. PMID 21369362
- [Background] Mazzucchelli T, Kane R, Rees CS. Behavioural activation treatments for depression in adults: A meta-analysis and review. Clin Psychol-Sci Pr 16(4): 383-411, 2009.
- [Background] McDonald S, Tate R, Togher L, Bornhofen C, Long E, Gertler P, Bowen R. Social skills treatment for people with severe, chronic acquired brain injuries: a multicenter trial. Arch Phys Med Rehabil. 2008 Sep;89(9):1648-59. doi: 10.1016/j.apmr.2008.02.029. PMID 18760150
- [Background] Medley AR, Powell T. Motivational Interviewing to promote self-awareness and engagement in rehabilitation following acquired brain injury: A conceptual review. Neuropsychol Rehabil. 2010 Aug;20(4):481-508. doi: 10.1080/09602010903529610. Epub 2010 Feb 1. PMID 20182952
- [Background] Oddy M, Cattran C, Wood R. The development of a measure of motivational changes following acquired brain injury. J Clin Exp Neuropsychol. 2008 Jul;30(5):568-75. doi: 10.1080/13803390701555598. PMID 18569252
- [Background] Richards DA, Ekers D, McMillan D, Taylor RS, Byford S, Warren FC, Barrett B, Farrand PA, Gilbody S, Kuyken W, O'Mahen H, Watkins ER, Wright KA, Hollon SD, Reed N, Rhodes S, Fletcher E, Finning K. Cost and Outcome of Behavioural Activation versus Cognitive Behavioural Therapy for Depression (COBRA): a randomised, controlled, non-inferiority trial. Lancet. 2016 Aug 27;388(10047):871-80. doi: 10.1016/S0140-6736(16)31140-0. Epub 2016 Jul 23. PMID 27461440
- [Background] Roozenbeek B, Maas AI, Menon DK. Changing patterns in the epidemiology of traumatic brain injury. Nat Rev Neurol. 2013 Apr;9(4):231-6. doi: 10.1038/nrneurol.2013.22. Epub 2013 Feb 26. PMID 23443846
- [Background] Teasell R, Bayona N, Marshall S, Cullen N, Bayley M, Chundamala J, Villamere J, Mackie D, Rees L, Hartridge C, Lippert C, Hilditch M, Welch-West P, Weiser M, Ferri C, McCabe P, McCormick A, Aubut JA, Comper P, Salter K, Van Reekum R, Collins D, Foley N, Nowak J, Jutai J, Speechley M, Hellings C, Tu L. A systematic review of the rehabilitation of moderate to severe acquired brain injuries. Brain Inj. 2007 Feb;21(2):107-12. doi: 10.1080/02699050701201524. PMID 17364527
- [Background] Turner-Stokes L. Evidence for the effectiveness of multi-disciplinary rehabilitation following acquired brain injury: a synthesis of two systematic approaches. J Rehabil Med. 2008 Oct;40(9):691-701. doi: 10.2340/16501977-0265. PMID 18843419
- [Background] Waldron B, Casserly LM, O'Sullivan C. Cognitive behavioural therapy for depression and anxiety in adults with acquired brain injury: what works for whom? Neuropsychol Rehabil. 2013;23(1):64-101. doi: 10.1080/09602011.2012.724196. Epub 2012 Nov 5. PMID 23121258
- [Background] Whelan-Goodinson R, Ponsford J, Johnston L, Grant F. Psychiatric disorders following traumatic brain injury: their nature and frequency. J Head Trauma Rehabil. 2009 Sep-Oct;24(5):324-32. doi: 10.1097/HTR.0b013e3181a712aa. PMID 19858966
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Derived] Kusec A, Murphy FC, Peers PV, Bennett R, Carmona E, Korbacz A, Lawrence C, Cameron E, Bateman A, Watson P, Allanson J, duToit P, Manly T. Mood, Activity Participation, and Leisure Engagement Satisfaction (MAPLES): results from a randomised controlled pilot feasibility trial for low mood in acquired brain injury. BMC Med. 2023 Nov 16;21(1):445. doi: 10.1186/s12916-023-03128-7. PMID 37974189
- [Derived] Kusec A, Murphy FC, Peers PV, Lawrence C, Cameron E, Morton C, Bateman A, Watson P, Manly T. Mood, Activity Participation, and Leisure Engagement Satisfaction (MAPLES): a randomised controlled pilot feasibility trial for low mood in acquired brain injury. Pilot Feasibility Stud. 2020 Sep 22;6:135. doi: 10.1186/s40814-020-00660-8. eCollection 2020. PMID 32974044

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT03874650/Prot_SAP_002.pdf